CLINICAL TRIAL: NCT01176123
Title: Comparing Telemedicine to In Person Delivery of Cognitive Behavioral Therapy for Trauma-Related Insomnia in Rural Veterans
Brief Title: Cognitive Behavioral Therapy for Trauma-Related Insomnia in Veterans
Acronym: CBT-I Telemed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast Louisiana Veterans Health Care System (U.S. Federal Agency)
Collaborators: VISN 16 Mental Illness Research, Education and Clinical Center (MIRECC) (Unknown)
Responsible Party: Principal Investigator, C Laurel Franklin, PhD, Staff Psychologist, Southeast Louisiana Veterans Health Care System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00366
Record Dates: First submitted 2010-08-04; First posted 2010-08-05 (Estimated); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: Cognitive behavioral therapy; Insomnia; Traumatic Stress
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-I in person (Active Comparator): Cognitive behavioral therapy for insomnia delivered in person
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia
- CBT-I via telephone therapy (Experimental): Cognitive behavioral therapy for insomnia delivered by telephone
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — Cognitive Behavioral Therapy for Insomnia

SUMMARY:
Understanding the effectiveness of Cognitive Behavioral Therapy for trauma-related insomnia (CBT-I) is important because sleep difficulties often persist after traditional post-trauma treatments are completed and other trauma-related symptoms have resolved. The objective of this study is to examine whether CBT-I will equivocally reduce problems falling and staying asleep (insomnia) related to military-related PTSD when administered in person versus through telephone therapy to veterans living in rural areas.

Rural populations are at a disadvantage in receiving treatment because of lack of access to healthcare services. Telemedicine uses technology (e.g., telephones) to provide distance counseling to the populations who lack access to health care. Thus, telephone-counseling strategies could provide broad access to interventions for management of trauma-related insomnia.

Veterans who live more than 30 miles from Veterans Affairs (VA) PTSD specialty services will be offered participation in this study. All veterans receive 6 weeks of individual CBT-I for trauma-related insomnia. Participants will be randomized to one of two treatment conditions: (1) CBT-I in person or (2) CBT-I via telemedicine (defined as receiving treatment by telephone). No changes will be made to the CBT-I, other than mode of delivery, for the telemedicine group.

Through this study the investigators hope to demonstrate the effectiveness of CBT-I for trauma-related insomnia can be delivered effectively to rural veterans in person and via telemedicine.

ELIGIBILITY:
Inclusion Criteria:

* Veterans living 30 or more miles from VA PTSD specialty services
* Diagnosis of PTSD or subthreshold PTSD symptoms
* Trauma-related insomnia

Exclusion Criteria:

* Primary sleep disorder other than insomnia(e.g., Restless Leg Syndrome)
* Psychosis
* Active alcohol dependence
* Active drug dependence

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-02-03 (Actual); Study Completion 2011-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurel Franklin, PhD, Principal Investigator — Southeast Louisiana Veterans Health Care System; Sheila Corrigan, PhD, Principal Investigator — Southeast Louisiana Veterans Health Care System
Locations (1):
- Southeast Louisiana Veterans Health Care System, New Orleans, Louisiana, United States